CLINICAL TRIAL: NCT02639195
Title: The Impact of Small Bowel Obstruction (SBO) on Quality of Life (QOL); the Efficacy of a Manual Physical Therapy to Improve QOL in Subjects With a History of SBO
Brief Title: The Impact of Small Bowel Obstruction (SBO) on Quality of Life (QOL)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Clear Passage Therapies, Inc (Industry)
Responsible Party: Principal Investigator, Lawrence Wurn, CEO, Clear Passage Therapies, Inc
Other Study IDs: SBO-C2015-005
Record Dates: First submitted 2015-12-21; First posted 2015-12-24 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Small Bowel Obstruction; Quality of Life; Bowel Obstruction
MeSH Terms: conditions — Intestinal Obstruction | interventions — Therapeutics; Musculoskeletal Manipulations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treatment, retrospective: Retrospective analysis on patients treated with manual physical therapy in quality of life outcomes as measured by pre and post treatment questionnaires. Chart review.
  Interventions: Other: Treatment
- Untreated control: Prospective data collection via questionnaire of subjects with a history of small bowel obstruction in an observational manner. No treatment is performed.

INTERVENTIONS:
Other: Treatment — Retrospective chart review of patients treated with manual therapy.
  Other Names: Manual Therapy
  Groups: Treatment, retrospective

SUMMARY:
This study has two segments the first is a chart and outcome assessment of patients treated at Clear Passage (CP) with a history of small bowel obstruction (SBO). These patients have completed multiple questionnaires as a standard of care for outcome monitoring in the clinic setting, no new data will be collected. The second segment is a prospective observational, online questionnaire based study of subjects with a history of SBO not treated at CP. Data on the impact of quality of life (QOL) over time of subjects not treated at CP will be assessed using the same questionnaire used as standard of care in the clinic twice, 90 days apart. This will be accomplished using the NIH Assessment Center, with subjects able to complete the questionnaires with ease via the internet. As this segment is observational, there is minimal risk to these subjects. The data obtained from the untreated subjects will allow for reporting of overall impact on QOL in this population, data that is not available, as well as provide a control group for assessment of improvement for interventions for SBO.

DETAILED DESCRIPTION:
This study has two segments the first is a chart and outcome assessment of patients treated at Clear Passage (CP) with a history of small bowel obstruction (SBO). These patients have completed multiple questionnaires as a standard of care for outcome monitoring in the clinic setting, no new data will be collected. The second segment is a prospective observational, online questionnaire based study of subjects with a history of SBO not treated at CP. Data on the impact of quality of life (QOL) over time of subjects not treated at CP will be assessed using the same questionnaire used as standard of care in the clinic twice, 90 days apart. This will be accomplished using the NIH Assessment Center, with subjects able to complete the questionnaires with ease via the Assessment Center. As this segment is observational, there is minimal risk to these subjects. The data obtained from the untreated subjects will allow for reporting of overall impact on QOL in this population, data that is not available, as well as provide a control group for assessment of improvement for interventions for SBO.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 90 years old
* Previous diagnosis of partial or total bowel obstruction in the last 2 years.
* Able to complete the questionnaire online via Assessment Center.

Exclusion Criteria:

* Currently pregnant
* Cancer within the last 10 years
* Chemotherapy or radiation treatments within the last 10 years
* Prior treatment at Clear Passage

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population with a history of a bowel obstruction in the last 2 years.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-04 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 90 days
  Questionnaire based study for QOL changes over 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Rice, PhD, Study Director — Clear Passage Therapies
Locations (1):
- Clear Passage Physical Therapy, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided